#### **Assent Form**

## **University of Minnesota**

### Assent to Participate in Research

Title of Research Study: Utilizing Senior Companions to Enhance Dementia Care

Services and Supports: R61 Phase

Researcher: Joseph Gaugler, Ph.D.

**Sponsors:** National Institute on Aging and National Institutes of Health

#### What is research?

Doctors and researchers are committed to your care and safety. There are important differences between research and treatment plans:

- The goal of research is to learn new things in order to help groups of people in the future. Researchers learn things by asking a question, making a plan, and testing it.
- The goal of treatment is to help you get better by using medication, therapy, surgery or other things that usually makes people feel better. Sometimes treatments help make you feel better or get rid of the condition completely. Doctors can make changes to your treatment plan as needed.

## Why am I being asked to take part in this research study?

A research study is usually done to find a better way to treat people or to understand how things work. You are being asked to take part in this research study because you or your loved one are interested in our research and thought that a Senior Companion could help you discuss your memory concerns and connect you to resources in the community.

## What should I know about being in a research study?

You do not have to be in this study if you do not want to do so. It is up to you if you want to participate. If you want to, talk to your caregiving loved one or your legally authorized representative about any questions or concerns you have about the study. You can choose not to take part now and change your mind later if you want. If you decide you do not want to be in this study, no one will be mad at you. You can ask all the questions you want before you decide.

## Why is this research being done?

This research is being done to test if Senior Companions can help you better address your memory concerns.

## How long will the research last?

I expect that you will be in this research study for one session that will last 4 months.

# What happens if I say "Yes, I want to be in this research"?

If you agree to join this study, you will be allowed to go on living your life as normal. You will be

1

#### **Assent Form**

asked to complete an initial, 1-month, and 3-month survey, and also complete a more open-ended, recorded interview of the telephone after the 3-month survey. During this time, your Senior Companion will visit and help you.

### What happens to the information collected for the research?

The researchers will share your information, including research study records, to only people who have a need to review this information. For example, sometimes researchers need to share information with the University or other people that work in research to make sure the researchers are following the rules.

#### What else do I need to know?

You have the right to choose not agree to participate in this research study for any reason. If you do not verbally agree, then you and/or your loved one cannot participate in this study.

#### Who can I talk to?

For questions about research appointments, the research study, research results, or other concerns, call the study team at:

Researcher Name: Joseph Gaugler, Ph.D Researcher Affiliation: University of

Minnesota

Phone Number: 612-626-2485 Email Address: gaug0015@umn.edu Study Staff: Katie Louwagie, DNP Position: Research Coordinator Phone

Number: 612-626-4776

Email Address: wocke007@umn.edu

This research has been reviewed and approved by an Institutional Review Board (IRB), a group of people that look at the research before it starts. This group is part of the Human Research Protection Program (HRPP). To share concerns privately with the HRPP about your research experience, call the Research Participants' Advocate Line at 612-625-1650 or go to https://research.umn.edu/units/hrpp/research-participants/questions-concerns.

You are encouraged to contact the HRPP if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide feedback about this research.

# **Assent Form**

| To be completed by person obtaining verbal assent from the participant: | | | |
|---|---|---|---|
| Care Recipient's/Participant's response: | □Yes | □No | |
| Participant's Name (printed) | | _ | |
| Name (printed) of Person Obtaining Assent | | | Date |
| Signature of Person Obtaining Assent | | | |